CLINICAL TRIAL: NCT02675543
Title: Vitreous Inflammation in Standard and Heavy Silicone Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Francesco Semeraro, To Compare Vitreous Inflammation in Standard Versus Heavy Silicone Oil, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitreo002
Record Dates: First submitted 2016-01-25; First posted 2016-02-05 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Vitreous Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard silicone oil (Experimental): after vitreous removal, the vitreous chamber was filled with standard silicone oil (PDMS)
  Interventions: Device: Vitreous Tamponade with Silicone Oil
- Heavy silicone oil (Experimental): after vitreous removal, the vitreous chamber was filled with heavy silicone oil (Densiron 68)
  Interventions: Device: Vitreous Tamponade with Silicone Oil

INTERVENTIONS:
Device: Vitreous Tamponade with Silicone Oil

SUMMARY:
The inflammatory response after prolonged retinal detachment and after vitreoretinal surgery has its apex in the development of PVR that occurs when retinal cells are exposed to the inflammatory milieu in the humor vitreous.

This situation is common in complicated retinal detachment, but is amplified after invasive surgery and by the use of intraocular tamponades that float over a subtle film of liquid where the inflammatory cytokines and growth factors reach the critical concentration over the inferior retina.

Many authors have noted that the heavy tamponade are more prone to cause intraocular inflammation compared to standard silicone oil, especially if they remain for several months in the eye.

The purpose of this study is to measure the vitreous concentration of some of the most important cytokines involved in the inflammatory vitreal response.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for vitrectomy

Exclusion Criteria:

* diabetic retinopathy
* uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual)

REFERENCES:
- [Derived] Schwartz SG, Flynn HW Jr, Wang X, Kuriyan AE, Abariga SA, Lee WH. Tamponade in surgery for retinal detachment associated with proliferative vitreoretinopathy. Cochrane Database Syst Rev. 2020 May 13;5(5):CD006126. doi: 10.1002/14651858.CD006126.pub4. PMID 32408387

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Silicone Oil: after vitreous removal, the vitreous chamber was filled with standard silicone oil (PDMS)
  Vitreous Tamponade with Silicone Oil
- Heavy Silicone Oil: after vitreous removal, the vitreous chamber was filled with heavy silicone oil (Densiron 68)
  Vitreous Tamponade with Silicone Oil
Period: Overall Study
Arm/Group | Standard Silicone Oil | Heavy Silicone Oil
Started | 15 | 20
Completed | 15 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Silicone Oil | Heavy Silicone Oil | Total
Number analyzed (Participants) | 15 | 20 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 16 | 26
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (12.8) | 62.3 (16.7) | 60.4 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 11 | 15 | 26
Region of Enrollment [Number; unit: participants]
  Italy | 15 | 20 | 35

OUTCOME MEASURES:

1. Primary Outcome: Vitreous Prostaglandin E2 Levels
Time Frame: intraoperarive
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Standard Silicone Oil | Heavy Silicone Oil
Number analyzed (Participants) | 15 | 20
pg/mL | 369.38 (209.7) | 869.16 (242.83)

ADVERSE EVENTS:
Arm/Group | Standard Silicone Oil | Heavy Silicone Oil
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/20
Other Adverse Events (participants affected / at risk) | 0/15 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No